CLINICAL TRIAL: NCT00527384
Title: Biomarker Signatures of Biological, Chemical, or Psychological Stress
Brief Title: Biomarker Analysis of Stress
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 16014-CP-001
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Sepsis
Keywords: Stress
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Physiological changes can occur from different types of stress as induced by an infection, an environmental toxicant exposure, or an emotional disturbance. The stress-induced effects can modify health by lessening defense mechanisms as maintained by the immune system. The ability of different forms of stress to alter physiological processes (body functions) will be assessed by monitoring the blood profile of cell numbers and functions as well as the plasma protein content. It is anticipated that the pattern of blood changes will reflect the types of stress and the degree to which body functions could be altered by the stress.

DETAILED DESCRIPTION:
Blood will be collected from patients with an ongoing infection that has lead to sepsis (systemic inflammation) as a index of major stress. The blood will be analyzed for the types of proteins that could alter immune system functions and affect organ functions, including cardiovascular effects due to blood vessel changes. This will be followed by analysis of stress effects on mice and mice that have been generated with human immune cells. The ability of stress to alter blood patterns will also be examined in mice with genetic modification of metallothionein expression, which is believe to influence oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Wadsworth Center with Sepsis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Lawrence, Ph.D., Principal Investigator — Wadsworth Center
Locations (1):
- Wadsworth Center, Albany, New York, United States